CLINICAL TRIAL: NCT03482024
Title: Pharmacokinetics of Tirzepatide Following Administration to Subjects With Impaired Renal Function
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Impaired Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17021; I8F-MC-GPGG (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-06-01

CONDITIONS: Renal Insufficiency; End Stage Renal Disease
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Tirzepatide - Control (Experimental): Group 1 - Tirzepatide 5 milligrams (mg) administered subcutaneously (SC) to healthy participants with normal renal function.
  Interventions: Drug: Tirzepatide
- Tirzepatide - Mild Renal Impairment (Experimental): Group 2 - Tirzepatide 5mg administered SC to participants with mild renal impairment.
  Interventions: Drug: Tirzepatide
- Tirzepatide - Moderate Renal Impairment (Experimental): Group 3 - Tirzepatide 5mg administered SC to participants with moderate renal impairment.
  Interventions: Drug: Tirzepatide
- Tirzepatide - Severe Renal Impairment (Experimental): Group 4 - Tirzepatide 5mg administered SC to participants with severe renal impairment.
  Interventions: Drug: Tirzepatide
- Tirzepatide - End Stage Renal Disease (ESRD) (Experimental): Group 5 - Tirzepatide 5mg administered SC to participants with ESRD.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC.
  Other Names: LY3298176

SUMMARY:
The purpose of this study is to assess how fast tirzepatide gets into the blood stream and how long it takes the body to remove it in participants with impaired kidney function compared to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* All Participants:

  * Women not of childbearing potential may participate and include those who are infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation), congenital anomaly such as mullerian agenesis; or postmenopausal
  * Are between the body mass index (BMI) of 19.0 and 40.0 kilograms per meter squared (kg/m²), inclusive, at screening
* Healthy Participants:

  -- Healthy males or females as determined by medical history, physical examination, and other screening procedures, with normal renal function, assessed by estimated glomerular filtration rate (eGFR) ≥90 milliliters per minute (mL/min) at screening
* Participants with Renal Impairment or ESRD:

  -- Males or females with stable mild to severe renal impairment, assessed by eGFR or with ESRD (having received hemodialysis for at least 3 months)
* Participants with Type 2 Diabetes Mellitus (T2DM) and Renal Impairment or ESRD:

  * Have T2DM controlled with diet or exercise alone or stable on metformin for at least 8 weeks
  * Taking stable doses of over-the-counter or prescription medications (eg, antihypertensive agents, aspirin, lipid-lowering agents) for treatment of concurrent medical conditions are permitted to participate providing they have been stable on their treatment regimen for at least 4 weeks
  * Have a hemoglobin A1c (HbA1c) ≥7.0% and ≤11.0% at screening

Exclusion Criteria:

* All Participants:

  * Women of childbearing potential
  * Have known allergies to tirzepatide or related compounds
  * Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2
  * Have serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2× the upper limit of normal (ULN) or total bilirubin (TBL) >1.5× ULN
  * Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis), elevation in serum amylase or lipase or GI disorder (eg, relevant esophageal reflux or gall bladder disease) or any GI disease which impacts gastric emptying (eg, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by glucagon-like peptide-1 (GLP-1) analogs or dipeptidyl peptidase IV (DPP-IV) inhibitors
* Participants with Renal Impairment or ESRD:

  * Have hemoglobin <8.5 grams per deciliter (g/dL) or significant active hematological disease from causes other than underlying renal disease.
  * Have used any drug indicated for medical care of the participant's renal impairment, which is not established in dose and administered for at least 7 days before LY3298176 administration
* Participants with T2DM and Renal Impairment or ESRD:

  * Have taken any glucose-lowering medications other than metformin, including insulin, in the past 3 months before screening
  * Have had more than 1 episode of severe hypoglycemia, as defined by the American Diabetes Association criteria, within 6 months before entry into the study or has a history of hypoglycemia unawareness or poor recognition of hypoglycemic symptoms

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Orange County Research Center, Tustin, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - High Point Clinical Trials Center, High Point, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Urva S, Quinlan T, Landry J, Martin J, Loghin C. Effects of Renal Impairment on the Pharmacokinetics of the Dual GIP and GLP-1 Receptor Agonist Tirzepatide. Clin Pharmacokinet. 2021 Aug;60(8):1049-1059. doi: 10.1007/s40262-021-01012-2. Epub 2021 Mar 29. PMID 33778934

RESULTS

PARTICIPANT FLOW:
Groups:
- Tirzepatide - Control: Participants received single dose of 5 milligram (mg) Tirzepatide by subcutaneous injection.
- Tirzepatide - Mild Renal Impairment; Tirzepatide - Moderate Renal Impairment; Tirzepatide - Severe Renal Impairment; Tirzepatide - End Stage Renal Disease (ESRD): Participants received single dose of 5mg Tirzepatide by subcutaneous injection.
Period: Overall Study
Arm/Group | Tirzepatide - Control | Tirzepatide - Mild Renal Impairment | Tirzepatide - Moderate Renal Impairment | Tirzepatide - Severe Renal Impairment | Tirzepatide - End Stage Renal Disease (ESRD)
Started | 14 | 8 | 8 | 7 | 8
Received At Least One Dose of Study Drug | 14 | 8 | 8 | 7 | 8
Completed | 13 | 8 | 8 | 7 | 8
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Tirzepatide - Control; Tirzepatide - Mild Renal Impairment; Tirzepatide - Moderate Renal Impairment; Tirzepatide - Severe Renal Impairment; Tirzepatide - End Stage Renal Disease (ESRD): Participants received single dose of 5mg Tirzepatide by subcutaneous injection.
- Total: Total of all reporting groups
Arm/Group | Tirzepatide - Control | Tirzepatide - Mild Renal Impairment | Tirzepatide - Moderate Renal Impairment | Tirzepatide - Severe Renal Impairment | Tirzepatide - End Stage Renal Disease (ESRD) | Total
Number analyzed (Participants) | 14 | 8 | 8 | 7 | 8 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (7.6) | 63.3 (6.6) | 68.8 (14.1) | 60.3 (9.3) | 52.9 (7.2) | 60.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 4 | 1 | 2 | 15
  Male | 9 | 5 | 4 | 6 | 6 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 3 | 4 | 0 | 14
  Not Hispanic or Latino | 12 | 3 | 5 | 3 | 8 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 2 | 3 | 1 | 8 | 21
  White | 7 | 6 | 3 | 6 | 0 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 8 | 8 | 7 | 8 | 45

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of Tirzepatide From Time Zero to Tlast (AUC[0-tlast])
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Time Zero to tlast (AUC[0-tlast]) of Tirzepatide was evaluated.
Time Frame: Predose, 8hours(h), 12h, 24h, 48h, 72h, 96h, 168h, 336h postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per Millilitre (ng*h/mL)
Arm/Group | Tirzepatide - Control | Tirzepatide - Mild Renal Impairment | Tirzepatide - Moderate Renal Impairment | Tirzepatide - Severe Renal Impairment | Tirzepatide - End Stage Renal Disease (ESRD)
Number analyzed (Participants) | 13 | 8 | 8 | 6 | 8
Nanogram*hour per Millilitre (ng*h/mL) | 78400 (24) | 81900 (36) | 98300 (32) | 81200 (9) | 88500 (14)

2. Primary Outcome: PK: Maximum Concentration of Tirzepatide
Description: Cmax is the maximum observed concentration of Tirzepatide.
Time Frame: Predose, 8hours(h), 12h, 24h, 48h, 72h, 96h, 168h, 336h postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per Millilitre (ng/mL)
Arm/Group | Tirzepatide - Control | Tirzepatide - Mild Renal Impairment | Tirzepatide - Moderate Renal Impairment | Tirzepatide - Severe Renal Impairment | Tirzepatide - End Stage Renal Disease (ESRD)
Number analyzed (Participants) | 13 | 8 | 8 | 6 | 8
Nanogram per Millilitre (ng/mL) | 339 (21) | 353 (42) | 369 (36) | 417 (11) | 347 (30)

3. Primary Outcome: PK: Area Under the Concentration Versus Time Curve (AUC) of Tirzepatide From Time Zero to Infinity (AUC[0-inf])
Description: Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC[0-inf]) of Tirzepatide was evaluated.
Time Frame: Predose, 8hours(h), 12h, 24h, 48h, 72h, 96h, 168h, 336h postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per Millilitre (ng*h/mL)
Arm/Group | Tirzepatide - Control | Tirzepatide - Mild Renal Impairment | Tirzepatide - Moderate Renal Impairment | Tirzepatide - Severe Renal Impairment | Tirzepatide - End Stage Renal Disease (ESRD)
Number analyzed (Participants) | 13 | 8 | 8 | 6 | 8
Nanogram*hour per Millilitre (ng*h/mL) | 80500 (25) | 84200 (37) | 10400 (32) | 83000 (10) | 93400 (12)

ADVERSE EVENTS:
Time Frame: Up to 28days
Groups:
- Tirzepatide - Control: Participants received single dose of 5 5mg Tirzepatide by subcutaneous injection.
Arm/Group | Tirzepatide - Control | Tirzepatide - Mild Renal Impairment | Tirzepatide - Moderate Renal Impairment | Tirzepatide - Severe Renal Impairment | Tirzepatide - End Stage Renal Disease (ESRD)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/8 | 0/8 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/8 | 0/8 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 1/14 | 4/8 | 3/8 | 3/7 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tirzepatide - Control (N=14) | Tirzepatide - Mild Renal Impairment (N=8) | Tirzepatide - Moderate Renal Impairment (N=8) | Tirzepatide - Severe Renal Impairment (N=7) | Tirzepatide - End Stage Renal Disease (ESRD) (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT03482024/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT03482024/SAP_001.pdf